CLINICAL TRIAL: NCT03754218
Title: Phase 1 Study of Human Amnion Membrane Powder for Enhanced Wound Healing
Brief Title: Amnion Wound Covering for Enhanced Wound Healing
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00054157
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-05

CONDITIONS: Burns; Wound of Skin; Skin Wound
Keywords: Human amnion membrane; Autologous skin graft; Scar Formation
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amnion membrane product treatment area (Experimental): The prepared amnion membrane powder will be directly applied to the prepared donor wound site (Site A). The wound will then be covered with the SOC dressing.
  Interventions: Drug: Amnion Membrane Powder; Procedure: SOC Wound Covering
- SOC Wound Covering treatment area (Active Comparator): The donor wound site (Site B) will be covered per SOC (Standard of care).
  Interventions: Procedure: SOC Wound Covering

INTERVENTIONS:
Drug: Amnion Membrane Powder — This sterilized product is composed of lyophilized, gamma-irradiated powder made from amniotic membrane for topical application with the purpose of enhanced wound healing.
  Arms: Amnion membrane product treatment area
Procedure: SOC Wound Covering — Institutional standard of care wound covering.

SUMMARY:
The purpose of this research study is to find our if human amnion membrane powder can be safely used as a covering for wounds and can improve the condition of skin graft donor sites. The amnion powder product is composed of "lyophilized" (freeze-dried), "gamma irradiation sterilized" (exposed to bacteria killing radiation) fragments of amniotic membrane.

DETAILED DESCRIPTION:
Extensive burns and full thickness skin wounds can be devastating to patients, even when treated with our current standard of care. There are an estimated 500,000 burns treated in the United States each year. Moreover, in the military environment, soldiers who suffer from extensive burn injuries on the battlefield may benefit from rapid treatments that result in complete closure and protection of the wounds. As such, there is a need for mobile platform technologies that allow fast treatment at the site where the injury occurred, or at the very least at the forward operating sites. This safety investigation of a human amnion membrane powder product for wound healing is a with-in patient-controlled study, enrolling 10 subjects undergoing donor skin graft harvest. The single-center study will include patients undergoing donor skin harvest such that two regions, of at least 25 cm2 and separated by at least a 5 cm gap, of donor site wounds in comparable skin locations, are available for covering with the amnion membrane product and the current institutional standard of care (SOC) covering. The proposed sterilized product is composed of lyophilized, gamma-irradiated powder made from amniotic membrane for topical application with the purpose of enhanced wound healing.

The primary objective of the study is to evaluate the safety of a human amnion membrane product intended for enhanced wound healing. The secondary objective is efficacy as evidenced by complete wound closure relative to standard of care (SOC) treatment in a similar wound on the same subject at donor sites created for skin grafts at 14 days and 28 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* The subject requires autologous primary skin graft with two donor sites in similar areas, each measuring at least 25 cm2 with the likely depth of 0.012 inches and separated by a 5 cm gap. It is preferable that the two sites be on right and left sides of the body, but it is not an exclusion if they must be on the same side.
* Eligible primary wound sites may be traumatic or chronic, and will be at least 50 cm2 (that will receive the donor graft) to allow assessment of two separate experimental donor sites of 25 cm2.
* The subject is between the ages of 18 and 85 years of age.
* The subject is willing to complete all follow-up evaluations required by the study protocol.
* The subject is to abstain from any other covering or treatment of the wound(s) for the duration of the study unless medically necessary.
* The subject agrees to abstain from enrollment in any other interventional clinical trial for the duration of the study.
* The subject and/or guardian is able to read and understand instructions and give informed, voluntary, written consent.
* The subject is able and willing to follow the protocol requirements

Exclusion Criteria:

* The subject's primary wound site is less than 50 cm2The subject's primary wound site is not deemed appropriate for skin graft based upon the investigator's clinical experience
* The subject has a microbiologically proven pre-existing local or systemic bacterial infection.
* The subject has been receiving a systemic antibiotic for more than 48 hours prior to grafting.
* Unstable cardiac disorders within the past 6 months including angina, abnormal ECG, history of cardiac arrest, surgery and/or other interventional procedure.
* Hepatic disease or altered liver function as defined by ALT or AST value >3 times the upper limit of normal and/or T. Bilirubin >1.5 mg/dL at screening
* Renal disease or altered renal function as defined by serum creatinine > 2 mg/dL at screening, or end-stage renal disease.
* Hemoglobin <10.0 or >19.0 g/dL
* Known coagulopathy or platelet disorder, or INR > 1.6 , PTT > 38 sec; PLT < 50,000 at screening
* The subject is known to have a pre-existing, chronic condition that, in the opinion of the Investigator, may interfere with wound healing including but not limited to: current malignancy, uncontrolled diabetes (HbA1c >8) or diabetic ulcers, autoimmune disease or other immunocompromised diseases, renal impairment or ESRD, liver disease, hematological

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Donor Site Wound Closure | Week 4
  Wound closure for both amnion membrane product and SOC will be defined as skin re-epithelization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart.

SECONDARY OUTCOMES:
Incidence of Donor Site Wound Healing | week 12
  Wound Healing for both amnion membrane product and SOC will be assessed clinically confirmed at two consecutive study visits 2 weeks apart.
Presence of infection | up to 26 Weeks
  The presence of infection will be evaluated in accordance with guidelines derived from Cutting and Harding using standard clinical measures.
Vancouver Scar Assessment Scale | up to 26 Weeks
  Scar formation will be evaluated the Vancouver Scar Assessment Scale.The scale is composed by the following Sub scales (minimum and maximum ranges in parenthesis): Pigmentation (0-2), Vascularity (0-3), Pliability (0-5), Height (0-3). Total score 0-13. Lower score denotes better outcomes for total range and subscales.
Presence of Dermatitis | Up to 26 Weeks
  Allergic Response to Human Amnion Membrane Product Covering will be assessed clinically by the presence of dermatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Molnar, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lesher AP, Curry RH, Evans J, Smith VA, Fitzgerald MT, Cina RA, Streck CJ, Hebra AV. Effectiveness of Biobrane for treatment of partial-thickness burns in children. J Pediatr Surg. 2011 Sep;46(9):1759-63. doi: 10.1016/j.jpedsurg.2011.03.070. PMID 21929986
- [Background] Rahmanian-Schwarz A, Beiderwieden A, Willkomm LM, Amr A, Schaller HE, Lotter O. A clinical evaluation of Biobrane((R)) and Suprathel((R)) in acute burns and reconstructive surgery. Burns. 2011 Dec;37(8):1343-8. doi: 10.1016/j.burns.2011.07.010. Epub 2011 Aug 17. PMID 21852044
- [Background] PIGEON J. Treatment of second-degree burns with amniotic membranes. Can Med Assoc J. 1960 Oct 15;83(16):844-5. No abstract available. PMID 13735672
- [Background] Faulk WP, Matthews R, Stevens PJ, Bennett JP, Burgos H, Hsi BL. Human amnion as an adjunct in wound healing. Lancet. 1980 May 31;1(8179):1156-8. doi: 10.1016/s0140-6736(80)91617-7. PMID 6155575
- [Background] Bose B. Burn wound dressing with human amniotic membrane. Ann R Coll Surg Engl. 1979 Nov;61(6):444-7. PMID 496235
- [Background] Koob TJ, Rennert R, Zabek N, Massee M, Lim JJ, Temenoff JS, Li WW, Gurtner G. Biological properties of dehydrated human amnion/chorion composite graft: implications for chronic wound healing. Int Wound J. 2013 Oct;10(5):493-500. doi: 10.1111/iwj.12140. Epub 2013 Aug 1. PMID 23902526
- [Background] Sawhney CP. Amniotic membrane as a biological dressing in the management of burns. Burns. 1989 Oct;15(5):339-42. doi: 10.1016/0305-4179(89)90015-6. PMID 2590408
- [Background] C. Ho, K. Tran, M. Hux, G. Sibbald, K. Campbell, Artificial skin grafts in chronic wound care: A meta-analysis of clinical efficacy and a review of cost-effectiveness, (2005).
- [Background] Thapliyal, G.K., Kumar, V. and Gour, S., Amniotic Membrane: An Innovative Material for Repair and Regeneration in Oral and Maxillofacial region-A Review. Rama University Journal & Dental Sciences, 3(2) (2016) 1-6.
- [Background] J.S. Davis, Skin transplantation, Johns Hopkins Hospital Reports 15 (1910) 307-96
- [Background] Pachigolla G, Prasher P, Di Pascuale MA, McCulley JP, McHenry JG, Mootha VV. Evaluation of the role of ProKera in the management of ocular surface and orbital disorders. Eye Contact Lens. 2009 Jul;35(4):172-5. doi: 10.1097/ICL.0b013e3181a66a12. PMID 19474753
- [Background] Honavar SG, Bansal AK, Sangwan VS, Rao GN. Amniotic membrane transplantation for ocular surface reconstruction in Stevens-Johnson syndrome. Ophthalmology. 2000 May;107(5):975-9. doi: 10.1016/s0161-6420(00)00026-9. PMID 10811093
- [Background] Mohammadi AA, Seyed Jafari SM, Kiasat M, Tavakkolian AR, Imani MT, Ayaz M, Tolide-ie HR. Effect of fresh human amniotic membrane dressing on graft take in patients with chronic burn wounds compared with conventional methods. Burns. 2013 Mar;39(2):349-53. doi: 10.1016/j.burns.2012.07.010. Epub 2012 Aug 27. PMID 22951345
- [Background] Branski LK, Herndon DN, Celis MM, Norbury WB, Masters OE, Jeschke MG. Amnion in the treatment of pediatric partial-thickness facial burns. Burns. 2008 May;34(3):393-9. doi: 10.1016/j.burns.2007.06.007. Epub 2007 Oct 24. PMID 17920202
- [Background] Ravishanker R, Bath AS, Roy R. "Amnion Bank"--the use of long term glycerol preserved amniotic membranes in the management of superficial and superficial partial thickness burns. Burns. 2003 Jun;29(4):369-74. doi: 10.1016/s0305-4179(02)00304-2. PMID 12781617
- [Background] Hermans MH. Preservation methods of allografts and their (lack of) influence on clinical results in partial thickness burns. Burns. 2011 Aug;37(5):873-81. doi: 10.1016/j.burns.2011.01.007. Epub 2011 Feb 25. PMID 21353745
- [Background] Fairbairn NG, Randolph MA, Redmond RW. The clinical applications of human amnion in plastic surgery. J Plast Reconstr Aesthet Surg. 2014 May;67(5):662-75. doi: 10.1016/j.bjps.2014.01.031. Epub 2014 Jan 31. PMID 24560801
- [Background] Lo K, Kohanim S, Trief D, Chodosh J. Role of amniotic membrane transplantation in acute chemical injury. Int Ophthalmol Clin. 2013 Fall;53(4):33-41. doi: 10.1097/IIO.0b013e31829ceec8. No abstract available. PMID 24088931
- [Background] Tseng SC, Prabhasawat P, Lee SH. Amniotic membrane transplantation for conjunctival surface reconstruction. Am J Ophthalmol. 1997 Dec;124(6):765-74. doi: 10.1016/s0002-9394(14)71693-9. PMID 9402822
- [Background] Ganatra MA. Amniotic membrane in surgery. J Pak Med Assoc. 2003 Jan;53(1):29-32. No abstract available. PMID 12666850
- [Background] Koziak A, Salagierski M, Marcheluk A, Szczesniewski R, Sosnowski M. Early experience in reconstruction of long ureteral strictures with allogenic amniotic membrane. Int J Urol. 2007 Jul;14(7):607-10. doi: 10.1111/j.1442-2042.2007.01781.x. PMID 17645603
- [Background] Tao H, Fan H. Implantation of amniotic membrane to reduce postlaminectomy epidural adhesions. Eur Spine J. 2009 Aug;18(8):1202-12. doi: 10.1007/s00586-009-1013-x. Epub 2009 Apr 30. PMID 19404691
- [Background] Chou CT, Lee C, Hwang JL. Amniotic membrane used for vulvar adhesion treatment. Arch Gynecol Obstet. 2001 Nov;265(4):223-4. doi: 10.1007/s004040000164. PMID 11789753
- [Background] Fetterolf DE, Snyder RJ. Scientific and clinical support for the use of dehydrated amniotic membrane in wound management. Wounds. 2012 Oct;24(10):299-307. PMID 25876055
- [Background] Zelen CM, Serena TE, Denoziere G, Fetterolf DE. A prospective randomised comparative parallel study of amniotic membrane wound graft in the management of diabetic foot ulcers. Int Wound J. 2013 Oct;10(5):502-7. doi: 10.1111/iwj.12097. Epub 2013 Jun 7. PMID 23742102
- [Background] Zelen CM. An evaluation of dehydrated human amniotic membrane allografts in patients with DFUs. J Wound Care. 2013 Jul;22(7):347-8, 350-1. doi: 10.12968/jowc.2013.22.7.347. PMID 24159656
- [Background] C.M. Zelen, T.E. Serena, D.E. Fetterolf, Dehydrated human amnion/chorion membrane allografts in patients with chronic diabetic foot ulcers: a long-term follow-up study, Wound Medicine 4 (2014) 1-4
- [Background] Forbes J, Fetterolf DE. Dehydrated amniotic membrane allografts for the treatment of chronic wounds: a case series. J Wound Care. 2012 Jun;21(6):290, 292, 294-6. doi: 10.12968/jowc.2012.21.6.290. PMID 22886294
- [Background] Sheikh ES, Sheikh ES, Fetterolf DE. Use of dehydrated human amniotic membrane allografts to promote healing in patients with refractory non healing wounds. Int Wound J. 2014 Dec;11(6):711-7. doi: 10.1111/iwj.12035. Epub 2013 Feb 15. PMID 23409746
- [Background] Bujang-Safawi E, Halim AS, Khoo TL, Dorai AA. Dried irradiated human amniotic membrane as a biological dressing for facial burns--a 7-year case series. Burns. 2010 Sep;36(6):876-82. doi: 10.1016/j.burns.2009.07.001. Epub 2010 Mar 16. PMID 20236771
- [Background] Subach BR, Copay AG. The use of a dehydrated amnion/chorion membrane allograft in patients who subsequently undergo reexploration after posterior lumbar instrumentation. Adv Orthop. 2015;2015:501202. doi: 10.1155/2015/501202. Epub 2015 Jan 13. PMID 25653880
- [Background] Kurd SK, Hoffstad OJ, Bilker WB, Margolis DJ. Evaluation of the use of prognostic information for the care of individuals with venous leg ulcers or diabetic neuropathic foot ulcers. Wound Repair Regen. 2009 May-Jun;17(3):318-25. doi: 10.1111/j.1524-475X.2009.00487.x. PMID 19660039
- [Background] Sen CK, Gordillo GM, Roy S, Kirsner R, Lambert L, Hunt TK, Gottrup F, Gurtner GC, Longaker MT. Human skin wounds: a major and snowballing threat to public health and the economy. Wound Repair Regen. 2009 Nov-Dec;17(6):763-71. doi: 10.1111/j.1524-475X.2009.00543.x. PMID 19903300
- [Background] Cherry DK, Hing E, Woodwell DA, Rechtsteiner EA. National Ambulatory Medical Care Survey: 2006 summary. Natl Health Stat Report. 2008 Aug 6;(3):1-39. PMID 18972720
- [Background] Pitts SR, Niska RW, Xu J, Burt CW. National Hospital Ambulatory Medical Care Survey: 2006 emergency department summary. Natl Health Stat Report. 2008 Aug 6;(7):1-38. PMID 18958996
- [Background] Miller SF, Bessey P, Lentz CW, Jeng JC, Schurr M, Browning S; ABA NBR Committee. National burn repository 2007 report: a synopsis of the 2007 call for data. J Burn Care Res. 2008 Nov-Dec;29(6):862-70; discussion 871. doi: 10.1097/BCR.0b013e31818cb046. No abstract available. PMID 18997556
- [Background] Cutting KF, Harding KG. Criteria for identifying wound infection. J Wound Care. 1994 Jun 2;3(4):198-201. doi: 10.12968/jowc.1994.3.4.198. PMID 27922298
- [Background] Baryza MJ, Baryza GA. The Vancouver Scar Scale: an administration tool and its interrater reliability. J Burn Care Rehabil. 1995 Sep-Oct;16(5):535-8. doi: 10.1097/00004630-199509000-00013. PMID 8537427
- [Background] Molnar JA, Lew WK, Rapp DA, Gordon ES, Voignier D, Rushing S, Willner W. Use of standardized, quantitative digital photography in a multicenter Web-based study. Eplasty. 2009;9:e4. Epub 2009 Jan 12. PMID 19212431
- [Background] Dornseifer U, Lonic D, Gerstung TI, Herter F, Fichter AM, Holm C, Schuster T, Ninkovic M. The ideal split-thickness skin graft donor-site dressing: a clinical comparative trial of a modified polyurethane dressing and aquacel. Plast Reconstr Surg. 2011 Oct;128(4):918-924. doi: 10.1097/PRS.0b013e3182268c02. PMID 21681125

DOCUMENTS (1):
  • Informed Consent Form (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT03754218/ICF_000.pdf